CLINICAL TRIAL: NCT02974166
Title: Analysis of the Effects of the Osteopathic Manipulative Treatment in Carriers of Temporomandibular Disorders: Randomized Clinical Trial
Brief Title: Analysis of the Effects of the Osteopathic Manipulative Treatment in Carriers of Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Osteopatia (Other)
Responsible Party: Principal Investigator, Thiago Boeira Susin, PT, DO, PT, DO, Instituto Brasileiro de Osteopatia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InstitutoBOsteopatia
Record Dates: First submitted 2016-11-16; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular Disorder; Osteopathic Manipulative Treatment; Rigid Splint; Speech Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Communication Disorders | interventions — Ibuprofen; Anti-Inflammatory Agents; cyclobenzaprine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Group (Active Comparator): Individuals with temporomandibular disorder were used rigid occlusal splints and medication (Ibuprofen and Cyclobenzaprine Hydrochloride) under the dentist professor supervision. Likewise, speech therapists performed assessments, measurements, massages, stretches and therapeutic exercises for head, neck and mouth regions during four weeks.
  Interventions: Other: Conventional Group; Drug: Ibuprofen; Drug: Cyclobenzaprine Hydrochloride
- Osteopathic Group (Experimental): Individuals with temporomandibular disorder received the same assistance of Conventional Group, cited above, plus the osteopathic care during 20 to 30 minutes once a week until the end of dental and speech therapy treatments (4 weeks).
  Interventions: Other: Osteopathic Group; Drug: Ibuprofen; Drug: Cyclobenzaprine Hydrochloride

INTERVENTIONS:
Other: Conventional Group — Rigid occlusal splints and medication (Ibuprofen and Cyclobenzaprine Hydrochloride) were made and prescribed under the dentist professor supervision. Likewise, speech therapists performed assessments, measurements, massages, stretches and therapeutic exercises for head, neck and mouth regions.
  Arms: Conventional Group
Other: Osteopathic Group — Same assistance of Conventional Group, cited above, plus the osteopathic care during 20 to 30 minutes once a week during four weeks. The osteopathic treatment consisted in an individualized assessment of mobility restrictions of myofascial tissues and joints and the application of smooth techniques such myofascial release, membranous strain and counterstrain, muscle energy, cranial and high velocity and low amplitude.
  Arms: Osteopathic Group
Drug: Ibuprofen — The medication was prescribed by the dentist as nonsteroidal anti-inflammatory drug if necessary.
  Other Names: anti-inflammatory drug
Drug: Cyclobenzaprine Hydrochloride — The medication was prescribed by the dentist as muscle relaxer if necessary.
  Other Names: muscle relaxer

SUMMARY:
The purpose of this study is to determine whether osteopathic manipulative treatment associated to Dentistry care and speech therapy improves pain and function in individuals with temporomandibular disorders.

DETAILED DESCRIPTION:
A standardized TMD examination was executed in all patients by a dentist following the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/ TMD) questionnaire, Axis I and II, portuguese version. The RDC/ TMD is compound by a 31 items questionnaire and a ten items clinical exam. All these items are related to patients symptoms and signs; to mandibular functional impairment; and social-demographics, social-economics, psychological e psychosocial data. The first part as Axis I tend to clinical assess and classify the TMD and the second, as Axis II propose a chronic pain score that could quantify the psychosocial impairment and present a subjects profile.

Others assessment instruments utilized on the research were the VAS consists in a 10 cm horizontal line with "no pain" on the left side and "worst pain" on right side, then the subjects were instructed to vertical risk the level of pain. The digital caliper with a 0,03 mm precision was used to measure the maximal mouth opening (MMO) as the maximal inter-incisal vertical distance of the incisors. The subjects were seated at 90° with neutral head position and solicited to open their mouths the maximum they can unassisted and without pain, maximum unassisted opening and maximum assisted opening. Also, a portable digital pressure algometer for measuring sensitivity to pressure before it became painful. The masseters and temporalis muscles trigger point location were used as reference to guarantee the reproducibility of the proceeding as well as to assess the always the same site. The statistical analysis was performed using the means comparisons for the parametric tests through Student T test and for the non-parametrical data, Wilcoxon. Also, it was made the descriptive statistical with frequencies analysis.

ELIGIBILITY:
Inclusion Criteria:

* subjects of both genders with TMD diagnosed and minimum pain intensity of 40 mm on a visual analogue scale (VAS) who need dental treatment.

Exclusion Criteria:

* continuous use of analgesic medication, mouth opening above 40 mm, presence of any other orofacial pain not related to TMD and being under orthodontic or TMD treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain assessed by visual analogue scale.

SECONDARY OUTCOMES:
(RDC/ TMD) Research Diagnostic Criteria for Temporomandibular Disorders | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thiago B Susin, Principal Investigator — IBO
Locations (1):
- Brazilian Institute of Osteopathy, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No